CLINICAL TRIAL: NCT00872664
Title: Skin and Serum Carotenoids in Preterm Infants Fed on a Formula Supplemented With Carotenoids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Abbott (Industry)
Responsible Party: Dr. Gary Chan, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 31886; ANUS 0805
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Retinopathy of Prematurity
Keywords: ROP; anti-oxidants; carotenoids
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Carotenoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- formula with added carotenoids (Active Comparator): Both arms are double-blinded. Infant will be assigned to receive preterm formula with added carotenoids. If infant is receiving human milk then the study formula will only be used as a supplement.
  Interventions: Dietary Supplement: carotenoids
- formula without added carotenoids (Active Comparator): Both arms are double-blinded. This arm will use preterm formula as it is currently available, which is without any carotenoids. If the infant is receiving human milk, then the formula will be used as a supplement as needed.
  Interventions: Dietary Supplement: carotenoids

INTERVENTIONS:
Dietary Supplement: carotenoids — beta-carotene, lycopene, lutein

SUMMARY:
The primary objectives of this study are to compare the serum and skin concentrations of beta-carotene, lutein, and lycopene in preterm infants fed preterm formulas with mixed carotenoids to serum concentrations in preterm infants fed preterm formulas with no added carotenoids and to human milk fed infants.

The secondary objective of this study is to evaluate the effects of dietary carotenoids on the developing eye. Stages and zones of retinopathy of prematurity (ROP), retinal function, and retinal characteristics will also be examined.

DETAILED DESCRIPTION:
Infants that are born prior to 37 weeks gestation often face complications resulting from their prematurity. Preterm infants are susceptible to morbidities that are not common in healthy term infants. Underdeveloped organs such as the lungs, eye, intestine, and brain can reveal conditions unique to prematurity: chronic lung disease, bronchopulmonary dysplasia (BPD), retinopathy of prematurity (ROP), necrotizing enterocolitis, intraventricular hemorrhage (IVH), etc. Infants in the Newborn Intensive Care Unit (NICU) have increased inflammation and oxidative stress in association with common diseases of prematurity and as well as the treatments used to combat their illnesses (Gitto et al 2004; Ochoa et al 2003; Saugstad 2003).

According to the National Eye Institute (U.S. National Institutes of Health), retinopathy of prematurity affects approximately 50% of preterm infants that are born weighing 1250 g or less. While 90% of infants with retinopathy of prematurity (ROP) experience the milder form of the disease, which requires little or no medical treatment, severe ROP can lead to serious visual impairments or even blindness. This condition is of particular interest since Hylander et al. (Hylander et al 2001) have reported that human milk feeding of preterm infants (<1500 g birth weight) has been associated with a lower incidence of ROP and this association was proposed to be driven by the antioxidant content of human milk. Human milk provides a variety of antioxidants to the breastfed infant, including the carotenoids lutein, zeaxanthin, lycopene, and beta-carotene. As discussed earlier, lutein and zeaxanthin are concentrated to the eye and are thought to provide protection against both light-induced and metabolic oxidative damage.

The retina and retinal vasculature are the last eye structures to develop in the human fetus/neonate. Eyes of children with a history of ROP are reported to have retinal thinning with diffuse hypopigmentation, mild linearization, or mild tortuosity of the major vessel branch, mottled pigmentation of the macula, and other peripheral retinal anomalies (Minicucci et al 1999). The lack of pigmentation in the retinal structure might be explained by the deficit of lutein acquired by the fetus (by placental transfer during late gestation) or by the neonate through the diet (by preterm infant formulas devoid of these carotenoids). Preterm infants are at a nutritional disadvantage at birth as they have been deprived of the period of maximal transfer of nutrients during the last few weeks of pregnancy. Blood levels of beta-carotene have been associated with gestational age (Ostrea et al 1986) and cord blood levels of beta-carotene (Herrera et al 2004; Kiely et al 1999; Yeum et al 1998), lutein (Kiely et al 1999), and lycopene (Herrera et al 2004; Kiely et al 1999) were reported to be significantly lower than maternal levels. Stores of fat-soluble antioxidant vitamins also could be compromised due to the minimal fat deposition in the preterm infant.

It is therefore reasonable to suggest that providing preterm infants with a milk-based ready-to-feed (RTF) preterm infant formula with DHA and ARA supplemented with carotenoids, which are found in human milk, would result in serum carotenoid levels more like the breastfed infant. Further, increased dietary carotenoid intake by preterm infants might decrease the prevalence of morbidities that are associated with prematurity, such as ROP, bronchopulmonary dysplasia (BPD), and intraventricular hemorrhage (IVH).

ELIGIBILITY:
Inclusion Criteria:

* Birth weight 500-1500 g.
* Less than 33 weeks gestational age (GA) at birth. Maternal dates will be used to estimate GA except in instances where a scan or the neonatologist's estimate differs by two weeks or more. In this instance, the scan or neonatologist's estimate of GA will be used. In the case where one neonatologist's estimate or scan confirms maternal dates and the other estimate does not confirm maternal dates, use the estimate of maternal dates.
* Randomization within 96 hours of initiation of enteral feeding of >/= 60mL/kg/d of HM or formula
* Formula fed infants' feeding consists of no more than 20% from human milk.
* Enteral feeding initiated by 21 days of life (date of birth is Day 0 of life).
* Parent/LAR agrees to allow infants to receive the assigned SSC Advance or NeoSure Advance formula in-hospital starting with the first enteral feed after randomization. If mother is providing breast milk, formula will only be given if there is not sufficient mother's milk.
* Parent/LAR signed the informed consent.
* SGA infants and infants with PDA are eligible to participate.
* Singleton or twin births only. For twins to be eligible, both must meet inclusion criteria.

Exclusion Criteria:

* Serious congenital abnormalities that may affect growth and development.
* Grade III or IV IVH.
* Maternal incapacity: including maternal cocaine or alcohol abuse during pregnancy or current, or if the mother or infant is currently receiving treatment consistent with HIV therapy.
* History of major surgery (including surgery for NEC).
* Asphyxia (hypoxia and ischemia) as evident by severe and permanent neurological damage.
* Confirmed NEC (modified Bell's stage II or III) or positive blood cultures at the time of randomization
* Infants who are enrolled in this clinical study should be excluded from participation in other concomitant studies. This exclusion criterion can be reviewed on a case-by-case basis. For example, infants will not normally be excluded if only demographic data are being collected or outcome measures on treatment modalities common to current clinical practice are being gathered.

Max Age: 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2009-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The primary objective is to compare the serum and skin levels of carotenoids in preterm infants fed formulas with mixed carotenoids to serum and skin levels in preterm infants fed formulas/human milk with no added carotenoids. | 3 years

SECONDARY OUTCOMES:
The secondary objective of this study is to evaluate the effects of dietary carotenoids on the developing eye. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Gary M Chan, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States